CLINICAL TRIAL: NCT00008840
Title: A Randomized, Open Label, Comparative, Multicenter Trial of Voriconazole Vs. AmBisome for Empirical Antifungal Therapy in Immunocompromised Patients With Persistent Fever and Neutropenia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: DMID MSG 42; 150-603
Record Dates: First submitted 2001-01-18; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of 2 drugs (AmBisome versus voriconazole) in treating fungal infections. Immunocompromised patients, especially those with persistent fever and neutropenia, are at a high risk of developing deeply invasive, life-threatening fungal infections with Candida, Aspergillus, and other opportunistic fungal pathogens. The risk of fungal infection increases in direct proportion with severity of neutropenia and duration of fever. Antifungal therapy, therefore, is an important step in the amelioration of fungal disease.

DETAILED DESCRIPTION:
Patients are first split into groups to receive either voriconazole or AmBisome. Both drugs are given through a vein (IV) for at least 3 days. At the conclusion of 3 days, the voriconazole patients are then switched to oral voriconazole. The AmBisome patients continue with IV AmBisome. Both groups continue treatment until blood counts increase and fever subsides.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are at least 12 years of age.
* Are hospitalized with low white blood cell counts.
* Have received at least 96 hours of IV antibiotics.
* Have an oral temperature (or equivalent) of 38.0 C (100.4 F) or greater within the 24 hours before the study starts.
* Are not pregnant or breast-feeding.
* Agree to use a barrier method of contraception (e.g., a condom) during the study

Exclusion Criteria:

You will not be eligible for this study if you:

* Have a serious fungal infection.
* Have a history of an allergic reaction to antifungal agents.
* Are taking certain medications which may interfere with the study drug.
* Are participating in a clinical trial of any investigational drug.
* Have previously participated in this trial.
* Have any conditions which could affect your safety, make evaluation of response difficult, or make it unlikely that you can complete the course of therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 866
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Ellen Bradley, Birmingham, Alabama, United States